CLINICAL TRIAL: NCT01611961
Title: A Phase I Study to Assess the Safety, Tolerability and Pharmacokinetics of Docetaxel Lipid Microsphere for Injection in Cancer Patients Receiving Chemotherapy
Brief Title: Docetaxel Lipid Microsphere (DT-LM) for Injection in Chemotherapy Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenyang Pharmaceutical University (Other)
Responsible Party: Principal Investigator, Shi Yuankai, Ph.D, the Director of Oncology Department, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYPHU-DT-LM-01
Record Dates: First submitted 2012-05-29; First posted 2012-06-05 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Advanced Cancer
Keywords: Docetaxel; Lipid Microsphere; Neoplasms; Antineoplastic Agents; Pharmacologic Actions; Therapeutic Uses
MeSH Terms: conditions — Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DT-LM (Experimental): Docetaxel Lipid Microsphere (DT-LM)
  Interventions: Drug: DT-LM
- Taxotere (Active Comparator): Commerical Product
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: DT-LM — Intravenous infusion, Upto 6 dose levels have been studied i.e. 45, 60, 75, 90 105,and 120 mg/m2, Every 3 weeks.
  Other Names: Docetaxel Lipid Microsphere
  Arms: DT-LM
Drug: docetaxel — Intravenous infusion, 3 dose levels：60, 75, and 90 mg/m2, Every 3 weeks
  Other Names: Taxotere
  Arms: Taxotere

SUMMARY:
Docetaxel Lipid Microsphere (DT-LM) is a novel proprietary delivery system of docetaxel developed by Shenyang Pharmaceutical University. In this Phase I study, the DT-LM was evaluated for the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) in patients with advance solid tumors. It was also evaluated for pharmacokinetic and anti-tumor effects of DT-LM compared to commerical docetaxel.

DETAILED DESCRIPTION:
Docetaxel (currently marketed as Taxotere®), given by intravenous or intraperitoneal injection, has contributed significantly to the treatment of a variety of malignancies, such as ovarian, breast, gastric, and non-small-cell lung cancer (NSCLC), as well as head and neck cancer and some other cancers. In the preclinical, DT-LM showed reduced toxicity (especially myelosuppression）and comparable therapeutic efficacy. In clinic, it is believed that DT-LM will offer fewer side effects to the patient at similar doses, and possibly greater effectiveness when used at higher doses. DT-LM could not only avoid the serious hypersensitivity reactions caused by Tween 80, but also be stable, safe and convenient for clinical administration.

This study is designed to determine the following:

* The maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of DT-LM.
* The pharmacokinetics of docetaxel following intravenous administration of DT-LM.
* Any anti-tumor effects of DT-LM.

Controlled trial is also carrying out to reveal the differences in safety, pharmacokinetics and pharmacodynamics between DT-LM and Taxotere.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and < 65, with ECOG performance status 0-1,and Life expectancy of more than 3 months.
2. Have advanced (local and/or metastatic) histologically documented cancer considered unresponsive to available conventional modalities or treatments.
3. Have recovered from acute toxicities of prior treatment:

   * 4 weeks must have elapsed since receiving any investigational agent.
   * 4 weeks must have elapsed since receiving any radiotherapy, or treatment with cytotoxic or biologic agents (≥6 weeks for mitomycin or nitrosoureas).
   * 4 weeks must have elapsed since any prior surgery.
4. Be in adequate condition as evidenced by the following clinical laboratory values:

   * Absolute neutrophil count (ANC) ≥1,500/mm3.
   * Platelets ≥ 80,000/mm3.
   * Hemoglobin ≥ 9.0 g/dL.
   * WBC ≥ 4,000/mm3.
   * Total bilirubin ≤ 2.5 x institutional upper limit normal (ULN).
   * Transaminases AST (SGOT) and ALT (SGPT) ≤ 1.5 times ULN or ≤ 5 times ULN (liver metastasis).
   * Serum creatinine ≤ 1.2 times ULN, blood urea nitrogen≤ 1.2 times ULN.
5. both female and male patients must use adequate methods of contraception.
6. Patient or legal representative must understand the investigational nature of this study and sign an Institutional Review Board (IRB)/Independent Ethics Committee approved written informed consent form prior to treatment.

Exclusion Criteria:

1. Intolerance to any antineoplastic agents belonging to the taxoid family.
2. having failed a docetaxel-containing regimen or Having known non-controllable hypersensitivity to docetaxel or lipid microsphere.
3. Active uncontrolled bleeding or bleeding diathesis (e.g., active peptic ulcer disease).
4. Unstable or uncontrolled cardiac disease or hypertension.
5. With other serious internal diseases, uncontrolled infection or uncontrolled diabetes.
6. With Symptomatic brain metastasis not controlled.
7. Having pre-existing clinically significant neuropathy (NCI CTCAE Grade ≥ 2 neuromotor or Grade ≥ 2 neurosensory) except for abnormalities due to cancer.
8. Currently receiving any other standard or investigational treatment for cancer or any other investigational agent for any indication.
9. Requiring immediate palliative treatment of any kind including surgery and/or radiotherapy.
10. Female patients who are pregnant or breast-feeding.
11. Unwilling or unable to follow protocol requirements.
12. With history of serious allergic or allergy.
13. Not fit for the clinical trial judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The safety and tolerability | one year
  This Phase I, open-label, control,dose-escalation study was designed to determine the maximum tolerated dose (MTD) of DT-LM in patients with advanced cancer. DT-LM was administered by intravenous infusion, over 1 hour, once every 21 days until occurrence of disease progression or toxicity requiring early treatment discontinuation. Dose escalation was not done until the safety and tolerability at a given dose level has been confirmed.

SECONDARY OUTCOMES:
Assessment of pharmacokinetics of DT-LM and Taxotere: AUC and Cmax | one year
  The patients were evaluated for pharmacokinetic profile of DT-LM and Taxotere upto 48 hours post treatment after cycle 1 and cycle 2,respectively.
Objective tumour response according to RECIST | one year
  The anti-tumor effects were evaluated after every two cycles of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xing Tang, Ph.D, Study Director — Shenyang Pharmaceutical University
Locations (1):
- Cancer Institute & Hospital, Chinese Academy of Medical Sciences, Beijing, China